CLINICAL TRIAL: NCT07038057
Title: Comparison of Short Peptide and Whole Protein Formula in the Early Enteral Nutrition of Patients With Sepsis: a Single-Center, Prospective, Randomized Controlled Study
Brief Title: Comparison of Short Peptide and Whole Protein Formula in the Early Enteral Nutrition of Patients With Sepsis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Ming Zhong, Doctor, Shanghai Zhongshan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B2025-213R
Record Dates: First submitted 2025-05-12; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Sepsis; Nutrition
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short peptide formula (Experimental): Within 48 hours of ICU admission, short-peptide-based enteral nutrition (Peptisorb) will be initiated. For patients with impaired swallowing or unconsciousness, a nasogastric tube will be placed. Feeding will start with low-calorie or trophic feeding, reaching 70% of the target energy and 1.2-1.5 g/kg/day of protein within 7 days. Due to significant individual variability in energy expenditure among sepsis patients, indirect calorimetry (IC) will be used to measure energy needs. If IC is unavailable, a weight-based formula (20-25 kcal/kg/day) will be applied. If patients remain in the ICU after 7 days, feeding will be gradually increased to full energy and protein targets as tolerated, followed by a transition to whole-protein nutrition.
  Interventions: Dietary Supplement: Short peptide enteral nutrition
- Whole protein formula (Active Comparator): Within 48 hours of ICU admission, whole-protein-based enteral nutrition (Nutrison) will be initiated, with the remaining protocol identical to the short-peptide group.
  Interventions: Dietary Supplement: Whole protein enteral nutrition

INTERVENTIONS:
Dietary Supplement: Short peptide enteral nutrition — Short peptide formula enteral nutrition was initiated within 48 hours after admission to the ICU. For patients with poor swallowing function or no consciousness, nasogastric tubes were placed. Starting from low-calorie or nourishing feeding, 70% of the target energy should be achieved within 7 days, and the protein should be 1.2-1.5 g/kg/d. Due to the large individual differences in energy expenditure among patients with sepsis, the indirect calorimetry (IC) method was used to determine energy expenditure. If the IC method is not feasible, the calculation formula based on body weight: 20-25 kcal/kg/d should be applied for calculation. If the patient is not transferred out of the ICU after 7 days, continue to gradually increase to the target energy and protein requirements under tolerable conditions, and gradually transition to whole protein nutrition after 7 days.
  Arms: Short peptide formula
Dietary Supplement: Whole protein enteral nutrition — The whole protein formula enteral nutrition was initiated within 48 hours of admission to the ICU, and the rest were same.
  Arms: Whole protein formula

SUMMARY:
To explore the effects of early enteral nutrition with short peptide formula on energy metabolism and clinical outcomes in patients with sepsis based on blood samples, clinical database, full-spectrum metabolomics test and imaging data, and to form a theoretical basis for optimizing the formula of early enteral nutrition in patients with sepsis.

DETAILED DESCRIPTION:
This study is a single-center prospective trial. Based on the annual patient volume, available human resources, and funding at our research center, the expert team determined a sample size of 80 cases, with 40 cases in the experimental group and 40 in the control group. Eligible participants will be randomized 1:1 via computer-generated randomization into two groups, receiving either a short-peptide-based enteral nutrition formula or a whole-protein-based enteral nutrition formula.

Short-peptide formula group:

Within 48 hours of ICU admission, short-peptide-based enteral nutrition (Peptisorb) will be initiated. For patients with impaired swallowing or unconsciousness, a nasogastric tube will be placed. Feeding will start with low-calorie or trophic feeding, reaching 70% of the target energy and 1.2-1.5 g/kg/day of protein within 7 days. Due to significant individual variability in energy expenditure among sepsis patients, indirect calorimetry (IC) will be used to measure energy needs. If IC is unavailable, a weight-based formula (20-25 kcal/kg/day) will be applied. If patients remain in the ICU after 7 days, feeding will be gradually increased to full energy and protein targets as tolerated, followed by a transition to whole-protein nutrition.

Whole-protein formula group:

Within 48 hours of ICU admission, whole-protein-based enteral nutrition (Nutrison) will be initiated, with the remaining protocol identical to the short-peptide group.

The study will assess changes in metabolomics after 7 days of early enteral nutrition with different protein formulations in sepsis patients, as well as differences in nutritional status, biochemical markers, and short- and long-term clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent has been signed
2. Aged from 18 to 80 years old
3. Within 24 hours after admission to ICU
4. Sepsis was diagnosed according to the 2016 International Sepsis 3.0 diagnostic criteria
5. Without gastrointestinal perforation, bleeding, obstruction and other contraindications to enteral nutrition
6. Expected ICU stay for more than 7 days

Exclusion Criteria:

1. Receiving palliative care or expected to die within 72 hours
2. Pregnant or breastfeeding
3. Use of high dose vasopressor maintenance (norepinephrine dosage > 0.5 μg/kg/min)
4. Requiring restricted protein intake or additional protein supplementation (e.g., patients with hepatic encephalopathy, severe renal insufficiency, severe burns, severe malnutrition, etc..)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-06-25 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Metabolomics changes form | On the 7th day after enrollment
  Key assessments include: ① Concentration changes of differential metabolites in core pathways (BCAA, SCFA, bile acid metabolism); ② Correlation between metabolite fluctuations and nutritional markers (albumin, prealbumin); ③ Predictive modeling linking metabolic signatures to clinical outcomes (infection rate, ICU LOS). The above data were all normalized and ultimately presented in the form of a heatmap.

SECONDARY OUTCOMES:
Daily average protein intake | 7 days
  Daily average protein intake, including EN, PN, IVAA, and measurable oral protein supplements; oral diets with unquantifiable protein content excluded (Unit: g).
Daily average energy intake | 7 days
  Daily average energy intake (Unit: g).
Energy adequacy rate | On the 3rd and 7th day after enrollment
  Energy adequacy rate on the 3rd and 7th day after enrollment (Unit: %).
Inflammatory markers | 7 days
  Including C-reactive protein (CRP) (Unit: mg/L), White blood cell count (WBC) (Unit: *10^9/L), and Neutrophil count (Neut#) (Unit: *10^9/L).
Nutritional status | 7 days
  Albumin (Alb) (Unit: g/L) and Pre-albumin (PA) (Unit: mg/L).
Liver function | 7 days
  Bilirubin (BIL) (Unit: μmol/L)
Renal function | 7 days
  Blood urea nitrogen (BUN) (Unit: mmol/L) and Serum creatinine (Cr) (Unit: umol/L).
Enteral nutritional tolerance rate | 7 days
  Manifestations of enteral nutrition intolerance:
  Gastric retention (gastric residual volume > 500 mL within 4 hours) Severe nausea or vomiting; Abdominal distension; Diarrhea (≥ 3 bowel movements per day with loose stools, Bristol Stool Scale type 5-7); Hematochezia leading to hemodynamic instability.
Skeletal muscle depletion condition | 7 days
  A single cross-sectional image at the L3 level was obtained via CT scan. Skeletal muscle was identified and quantified within the image using Hounsfield Unit (HU) thresholds of -29 to +150. The total muscle area at this level was calculated using ImageJ image analysis software. After normalization by the square of height (m²), the third lumbar skeletal muscle index (L3-SMI) was derived.
Days of ventilator use | 28 days
28-day all-cause mortality rate | 28 days
All-cause mortality at 90 days | 90 days

IPD SHARING:
Plan to Share IPD: No